CLINICAL TRIAL: NCT02274727
Title: Biomarker Signature of Stroke Aetiology Study: The BIOSIGNAL-Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Mira Katan, Principal Investigator, University of Zurich
Other Study IDs: 2014-001
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Stroke, Acute
Keywords: Biomarker; Stroke; Etiology; Outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The three-year cumulative risk of a recurrent stroke, dependent on aetiology, is up to 25 per cent. At present, preventing recurrence relies on a broad approach to reduce risk factors associated with atherosclerosis, heart disease and metabolic disorders. However, more specific interventions, such as anticoagulation and surgery or stenting, need aetiologic information. BIOSIGNAL aims to determine where the most promising candidate biomarkers can help identify stroke aetiology and also predict overall MACE, including specifically recurrent stroke. In addition, the insights gained into the processes underlying different stroke subtypes may lead to more targeted diagnostic tools.

DETAILED DESCRIPTION:
Objectives and specific aims:

The investigators propose to prospectively evaluate the predictive value of the most promising blood bio-markers to identify treatable stroke etiologies on admission and risk of MACE and its components in consecutive ischemic stroke patients enrolled by several centers in Europe.

The clinical endpoints of the study are 1) recurrent cerebrovascular events (ischemic stroke and / or transient ischemic attack (TIA)) and major cardiac events (MACE) within one year after the index stroke and after 3-5 years of follow up (2021) 2) all types of atrial fibrillation (AF) detected on admission or by prolonged ambulatory cardiac rhythm monitors during the follow up period 3) presence of cerebrovascular atherosclerosis detected by ultrasound investigations and 4) overall mortality, functional outcome, cognitive impairment, occurrence of epilepsy, and newly diagnosed cancer, according to data collected in telephonic interviews in 2021 (only in Zurich and Basel) with the patients enrolled between 2014-2017.

Aim 1: To determine whether the proposed and novel biomarkers independently predict recurrent stroke and a composite outcome consisting of recurrent cerebrovascular event (ischemic stroke (AIS), intracranial hemorrhage (ICH) or transient ischemic attack (TIA), as well as myocardial infarction (MI), cardiovascular death (CVD)). i.e. major adverse cardiac events (MACE) among all patients. Hypothesis 1: Elevated levels of one or more of the proposed and novel biomarkers will independently predict MACE and its components during trial follow-up, assessed by structured interviews, as well as chart reviews 90 days, 1 year after the index stroke as well as in 2021 (only in Zurich and Basel).

Aim 2: To determine whether CE biomarkers are associated with atrial fibrillation among all patients. Hypothesis 2: Baseline values of one or more of the CE biomarkers will be independently associated with AF, including history of AF, AF detection at baseline, or AF detected during the follow up period by prolonged (at least 7-day) ambulatory cardiac rhythm monitors and structured interviews as well as chart reviews 90 days, 1 year after the index stroke as well as in 2021 (only in Zurich and Basel).

Aim 3: To determine whether LAA biomarkers are associated with a) the presence of cerebrovascular atherosclerosis among all patients. Hypothesis 3: Baseline values of one or more of LAA biomarkers will be independently associated with the presence of extra and intracranial atherosclerosis among patients with ischemic stroke.

Exploratory Aim 4: To determine whether the proposed and novel biomarkers will predict a) occurrence of epileptic seizures and diagnosis of epilepsy b) newly diagnosed cancer, c) functional outcome and cognitive impairment. Hypothesis 4: Baseline values of one or more of the proposed and potentially novel biomarkers will independently predict a) occurrence of epileptic seizures and the diagnosis of epilepsy b)occurrence of newly diagnosed cancer c) functional outcome and cognitive impairment assessed by a follow up structured telephone interview performed in 2021 with the patients enrolled between 2014-2017 (only in Zurich and Basel).

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, and Good Clinical Practice (GCP) guidelines as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients (above the age of 18) who are admitted with a suspected ischemic stroke within 24 hours of symptom onset are eligible.

Ischemic stroke is defined as an acute localized ischemic lesion in the brain not attributable to central nervous system infection, tumor, demyelinating, or degenerative neurologic diseases due to an occlusive vascular disorder.

Detailed Inclusion Criteria:

1. Rapid onset of a focal neurologic deficit, with signs or symptoms persisting beyond 24 hours & NOT associated with:

   * infection
   * trauma
   * tumor of the brain
   * severe metabolic disorders
   * chronic degenerative neurologic disease
2. The development of an acute focal neurologic deficit persisting >24 hours in conjunction with brain imaging consistent with acute ischemic stroke.

The CT or MRI may either show a new infarct or no change from the study performed at entry, i.e. the diagnosis is clinical and does not require CT/MRI confirmation. Secondary hemorrhagic infarction is permissible.

Exclusion Criteria:

1. Hemorrhagic stroke
2. All patients discharged from the hospital with a diagnosis different from ischemic stroke (i.e. stroke mimics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The BIOSIGNAL study will be a prospective observational multicenter cohort study to evaluate selected CE and LAA blood biomarkers in patients with incident ischemic stroke. We will consecutively recruit patients over a planned time period of two years. All participants will be followed for 1 year.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2014-09; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite of Major adverse cardiac events (MACE) | Within 1 year after the index event. In Zurich and Basel also in 2021
  Recurrent cerebrovascular events (ischemic stroke (AIS), intracranial hemorrhage (ICH) or transient ischemic attack (TIA)), as well as myocardial infarction (MI), cardiovascular death (CVD). i.e. major adverse cardiac events (MACE)

SECONDARY OUTCOMES:
Single components and combinations of MACE | Within one year after the index stroke
  Recurrent cerebrovascular events (ischemic stroke (AIS), intracranial hemorrhage (ICH) or transient ischemic attack (TIA)), myocardial infarction (MI) or cardiovascular death (CVD)
Stroke aetiology | During first hospitalisation (cross-sectional analysis, up to 14 days)
  According to TOAST and SS TOAST criteria
History of AF | Diagnosed befor the stroke
  Assessed by chart review and taking the patients history
Newly Atrial Fibrillation (AF) | On admission and during a one year of follow-up by PCM. In Zurich and Basel also in 2021
  Newly diagnosed atrial fibrillation in patients with no history of AF
The presence of cerebrovascular atherosclerosis among all patients. | During first hospitalisation (cross-sectional analysis, up to 14 days)
  Assessed by duplex sonography.

OTHER OUTCOMES:
Functional outcome | Within 3 month after the index stroke and at one year. In Zurich and Basel also in 2021
  Assessed by the modified Rankin scale (mRS)
Occurrence of epileptic seizures and the diagnosis of epilepsy | During 2021 (only in Zurich and Basel)
  According to the medical history reported by patient and a questionnaire
Ooccurrence of newly diagnosed cancer | During 2021 (only in Zurich and Basel)
  According to the medical history reported by patient
Cognitive impairment | During 2021 (only in Zurich and Basel)
  Assessed by the Telephone Interview for Cognitive Status (TICS) Questionnaire
Mortality | Within 1 year after the index event. In Zurich and Basel also in 2021
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Mira Katan, MD, MS, Principal Investigator — Name: Mira Katan, MD, Msc
Locations (9):
- University Hospital of Frankfurt, Frankfurt am Main, Germany
- Larissa University Hospital of Thessaly, Larissa, Greece
- Universitiy Hospital Vall d'Hebron, Barcelona, Spain
- Switzerland (6):
  - Kantonsspital Aarau, Department of Neurology, Aarau, Canton of Aargau
  - University Hospital of Basel, Basel
  - University Hospital of Bern/Inselspital, Bern
  - Stroke Center ; Neurocentro(EOC) della Svizzera Italiana, Lugano
  - Stroke Center, Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital of Zurich, Department of Neurology, Zurich

REFERENCES:
- [Derived] Cameron AC, Arnold M, Katsas G, Yang J, Quinn TJ, Abdul-Rahim AH, Campbell R, Docherty K, De Marchis GM, Arnold M, Kahles T, Nedeltchev K, Cereda CW, Kagi G, Bustamante A, Montaner J, Ntaios G, Foerch C, Spanaus K, Eckardstein AV, Dawson J, Katan M. Natriuretic Peptides to Classify Risk of Atrial Fibrillation Detection After Stroke: Analysis of the BIOSIGNAL and PRECISE Cohort Studies. Neurology. 2024 Aug 13;103(3):e209625. doi: 10.1212/WNL.0000000000209625. Epub 2024 Jul 1. PMID 38950311
- [Derived] Schweizer J, Arnold M, Konig IR, Bicvic A, Westphal LP, Schutz V, Inauen C, Scherrer N, Luft A, Galovic M, Ferreira Atuesta C, Pokorny T, Arnold M, Fischer U, Bonati LH, De Marchis GM, Kahles T, Nedeltchev K, Cereda CW, Kagi G, Bustamante A, Montaner J, Ntaios G, Sagris D, Foerch C, Spanaus K, von Eckardstein A, Katan M. Measurement of Midregional Pro-Atrial Natriuretic Peptide to Discover Atrial Fibrillation in Patients With Ischemic Stroke. J Am Coll Cardiol. 2022 Apr 12;79(14):1369-1381. doi: 10.1016/j.jacc.2022.01.042. PMID 35393018